CLINICAL TRIAL: NCT02695004
Title: Randomized, Double-blind, Placebo-controlled, Single Ascending Dose Phase 1 Clinical Trial to Evaluate Safety, Tolerability and Pharmacokinetics of DKF-310 Intramuscular Injection in Healthy Male Volunteers
Brief Title: Safety, Tolerability and Pharmacokinetics of DKF-310 ( (Donepezil).
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Dongkook Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: DKF-310-P1
Record Dates: First submitted 2016-02-18; First posted 2016-03-01 (Estimated); Last update posted 2020-04-06 (Actual); Status verified 2016-02

CONDITIONS: Alzheimer's Disease
MeSH Terms: conditions — Alzheimer Disease | interventions — Donepezil

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- Donepezil 35 mg (Experimental): Donepezil 35 mg or placebo
  Interventions: Drug: DKF-310; Drug: Placebo
- Donepezil 70 mg (Experimental): Donepezil 70 mg or placebo
  Interventions: Drug: DKF-310; Drug: Placebo
- Donepezil140 mg (Experimental): Donepezil 140 mg or placebo
  Interventions: Drug: DKF-310; Drug: Placebo
- Donepezil 210 mg (Experimental): Donepezil 210 mg or placebo
  Interventions: Drug: DKF-310; Drug: Placebo
- Donepezil 280 mg (Experimental): Donepezil 280 mg or placebo
  Interventions: Drug: DKF-310; Drug: Placebo

INTERVENTIONS:
Drug: DKF-310
  Other Names: Donepezil
Drug: Placebo

SUMMARY:
This is a study to evaluate safety, tolerability and PK of DKF-310 IM injection in healthy male volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Men aged 19 to 50 years
* Body weight 55 to 90 kg and BMI 18.0 to 27.0
* Voluntarily signed the informed consent form
* Eligible according to the screening test results
* Available to follow up after drop-out

Exclusion Criteria:

* Clinically significant disorders or a medical history of hepatic, renal, neurological, respiratory, endocrine, hemato-oncologic, cardiovascular, urological and psychiatric diseases
* Hypersensitivity to donepezil, piperidine derivatives and other drugs
* SBP <100 mmHg or >150 mmHg, or DBP <60 mmHg or >100 mmHg
* Skin and muscle disorders or history of surgery at the injection site
* AST or ALT >1.5xULN; QT/QTcB interval >450 ms
* History or positive result of drug abuse
* Prescribed drugs or herbal medicines within 2 weeks, over-the-counter drugs or vitamins within 1 week
* Participated in other clinical trials within 3 months
* Donated whole blood within 2 months or apheresis within 1 month, or transfusion within 1 month
* Alcohol consumption >21 units/week
* Smoked >10 cigarettes/day within 3 months
* Caffeine-containing foods
* Not eligible due to other reasons at the investigator's discretion

Ages: 19 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 44 (Actual)
Dates: Start 2016-02; Primary Completion 2017-03 (Actual); Study Completion 2017-03 (Actual)

PRIMARY OUTCOMES:
AUC | 1056h
  0, 0.5, 1, 2, 4, 6, 8, 12, 24, 48, 72, 96, 120, 168, 240, 312, 360, 408, 432, 456, 480, 504, 528, 552, 600, 720, 816, 888, 960, 1056h
Cmax | 1056h
  0, 0.5, 1, 2, 4, 6, 8, 12, 24, 48, 72, 96, 120, 168, 240, 312, 360, 408, 432, 456, 480, 504, 528, 552, 600, 720, 816, 888, 960, 1056h

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National Univ. Bundang Hospital, Seongnam, South Korea

IPD SHARING:
Plan to Share IPD: No